CLINICAL TRIAL: NCT06945484
Title: PILOT for The Precision Exercise Regimen for Cancer Care (PERCC) Study
Acronym: PILOT PERCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI162865
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage II; NSCLC, Stage III
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Precision Exercise Regimen for Cancer Care (PERCC) (Experimental): Participants will engage in PERCC starting at least two weeks prior to receiving their first neoadjuvant treatment for lung cancer and continuing until two months after receiving surgical treatment.
  Interventions: Other: Precision Exercise Regimen for Cancer Care (PERCC)

INTERVENTIONS:
Other: Precision Exercise Regimen for Cancer Care (PERCC) — PERCC has exercise modes including basic transfer and calisthenics mobility, aerobic, and resistance exercises, and will be performed in various postures (supine, sitting, standing, and walking) with variable challenges (level walking, bending, inclines, steps, and squatting). Each participant will complete one supervised, home-based exercise training session per week, delivered through telehealth, that will focus on the resistance exercise prescription. Other unsupervised exercise training sessions will focus on the aerobic exercise prescription and will be completed individually

SUMMARY:
This study is designed to evaluate whether a precision exercise regimen is feasible to implement within cancer populations, specifically stage II-III primary lung cancer patients receiving multimodal therapy, and delivered through telehealth.

DETAILED DESCRIPTION:
This is a pilot study evaluating the feasibility of the Precision Exercise Regimen for Cancer Care (PERCC) intervention in stage II and stage III Non-Small Cell Lung Cancer (NSCLC) patients receiving multimodal therapy at the Huntsman Cancer Institute (HCI) at the University of Utah. Eligible patients will begin the intervention at the pre-treatment clinic visit and continue until approximately two months post-surgery.

The PERCC intervention is a virtually supervised home-based exercise program. Participants will engage in exercise starting at least two weeks before receiving their first neoadjuvant treatment for lung cancer and continuing until two months after receiving surgical treatment. The exercise modes will include basic transfer and calisthenics mobility, aerobic, and resistance exercises and will be performed in various postures (supine, sitting, standing, and walking) with variable challenges (level walking, bending, inclines, steps, and squatting).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older at time of diagnosis
* Patient diagnosed with stage II and III non-small cell lung cancer (NSCLC)
* Patient receives either neoadjuvant chemotherapy or immunotherapy and surgery
* Patient able to follow direction and complete questionnaires in English or Spanish
* Patient agrees to complete the PERCC intervention

Exclusion Criteria:

* Morbidly obese (BMI >40 kg/m2 ) or anorexic (BMI <17.5 kg/m2 )
* Abnormalities on screening physical exam per study physicians or physical therapist to contraindicate participation in exercise program compliance
* Alcohol or drug abuse, significant mental or emotional problems that would interfere with compliance (assessed by NCCN Distress Thermometer)
* Patient scheduled to receive single modality cancer treatment (unimodal therapy), scheduled to begin treatment within 2 weeks of the pre-treatment clinic visit, or for whom treatment has already started

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment and Retention | up to two months post-surgery
  Feasibility of the PERCC intervention will be evaluated by our ability to recruit and retain the needed number of patients with 80% exercise intervention attendance.

SECONDARY OUTCOMES:
Feasibility - Safety | up to two months post-surgery
  The feasibility of the PERCC intervention will be evaluated based on participant safety.
  This outcome measure will assess the safety and tolerability of the study treatment.
  The severity of AEs will be assessed using CTCAE v5.0 criteria, a 1-5 scale with higher numbers indicating greater severity. Grade 1 indicates "mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated" and Grade 5 indicates "death related to AE".
  Subjects will be monitored for adverse events from the start of treatment until two months post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Ulrich, MS, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (2):
- United States (2):
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2016. CA Cancer J Clin. 2016 Jan-Feb;66(1):7-30. doi: 10.3322/caac.21332. Epub 2016 Jan 7. PMID 26742998
- [Background] Ettinger DS, Wood DE, Aggarwal C, Aisner DL, Akerley W, Bauman JR, Bharat A, Bruno DS, Chang JY, Chirieac LR, D'Amico TA, Dilling TJ, Dobelbower M, Gettinger S, Govindan R, Gubens MA, Hennon M, Horn L, Lackner RP, Lanuti M, Leal TA, Lin J, Loo BW Jr, Martins RG, Otterson GA, Patel SP, Reckamp KL, Riely GJ, Schild SE, Shapiro TA, Stevenson J, Swanson SJ, Tauer KW, Yang SC, Gregory K; OCN; Hughes M. NCCN Guidelines Insights: Non-Small Cell Lung Cancer, Version 1.2020. J Natl Compr Canc Netw. 2019 Dec;17(12):1464-1472. doi: 10.6004/jnccn.2019.0059. PMID 31805526
- [Background] Tchelebi LT, Shen B, Wang M, Potters L, Herman J, Boffa D, Segel JE, Park HS, Zaorsky NG. Nonadherence to Multimodality Cancer Treatment Guidelines in the United States. Adv Radiat Oncol. 2022 Mar 8;7(5):100938. doi: 10.1016/j.adro.2022.100938. eCollection 2022 Sep-Oct. PMID 35469182
- [Background] Gao SJ, Corso CD, Wang EH, Blasberg JD, Detterbeck FC, Boffa DJ, Decker RH, Kim AW. Timing of Surgery after Neoadjuvant Chemoradiation in Locally Advanced Non-Small Cell Lung Cancer. J Thorac Oncol. 2017 Feb;12(2):314-322. doi: 10.1016/j.jtho.2016.09.122. Epub 2016 Oct 5. PMID 27720827
- [Background] Hanna TP, King WD, Thibodeau S, Jalink M, Paulin GA, Harvey-Jones E, O'Sullivan DE, Booth CM, Sullivan R, Aggarwal A. Mortality due to cancer treatment delay: systematic review and meta-analysis. BMJ. 2020 Nov 4;371:m4087. doi: 10.1136/bmj.m4087. PMID 33148535
- [Background] Yalman D. Invited Editorial on "the timing of surgery after neoadjuvant chemoradiation in locally advanced non-small cell lung cancer". J Thorac Dis. 2017 Mar;9(3):E299-E300. doi: 10.21037/jtd.2017.02.98. No abstract available. PMID 28449527